CLINICAL TRIAL: NCT05845554
Title: Application of Chromosomal Instability and Metagenomic Detection in Early Diagnosis of Biliary Tract Carcinoma in Bile
Brief Title: Application of Chromosomal Instability in Early Diagnosis of Biliary Tract Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Collaborators: Taizhou First People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Fabiao zhang, department director, Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Other Study IDs: BileCAD-330
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Biliary Tract Carcinoma
Keywords: Biliary Tract Carcinoma; chromosomal instability
MeSH Terms: conditions — Chromosomal Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from cast-off cells in bile sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biliary tract carcinoma patients: Biliary tract carcinoma patients will be the experimental group to determine the sensitivity of BileCAD analysis.
  Interventions: Diagnostic Test: The extracted DNA from bile samples will be analyzed by BileCAD to determine the level of CIN.
- Non-cancer participants Patients: Non-cancer participants Patients being treated for other diseases but without any tumor will provide a negative control to provide data for determining the specificity of BileCAD analysis.
  Interventions: Diagnostic Test: The extracted DNA from bile samples will be analyzed by BileCAD to determine the level of CIN.

INTERVENTIONS:
Diagnostic Test: The extracted DNA from bile samples will be analyzed by BileCAD to determine the level of CIN. — The extracted gDNA from bile sample will be analyzed by BileCAD to determine the level of CINs.

SUMMARY:
Chromosomal instability (CIN) refers to ongoing chromosome segregation errors throughout consecutive cell divisions. CIN is a hallmark of human cancer, and it is associated with poor prognosis, metastasis, and therapeutic resistance. Analyzing CIN of the DNA extracted from cast-off cells in bile samples seems a promising method for diagnosing, monitoring, and predicting the prognosis of biliary tract carcinoma patients. CIN can be assessed using experimental techniques such as bulk DNA sequencing, fluorescence in situ hybridization (FISH), or conventional karyotyping. However, these techniques are either time-consuming or non-specific. The investigators here intend to study whether a new method named Bile Ultrasensitive Chromosomal Aneuploidy Detection (BileCAD), which is based on low-coverage whole-genome sequencing, can be used to analyze CIN and microbial infection analysis thus help diagnosing and treating biliary tract carcinoma patients.

DETAILED DESCRIPTION:
Biliary tract carcinoma account for about 3% of all digestive system tumors, with potential high metastasis and invasion ability. Their early clinical symptoms lack specificity, and they are often found in late stage with poor prognosis. CIN results from errors in chromosome segregation during mitosis, leading to structural and numerical chromosomal abnormalities. It will generate genomic heterogeneity that acts as a substrate for natural selection. Furthermore, it is proved that tumors with aneuploidies and polyploidy resulting from whole-genome doubling are related with metastasis, treatment resistance, and decreased overall survival. It is estimated that 60%-80% of human tumors exhibit chromosomal abnormalities suggestive of CIN. CIN positively correlates with tumor stage and is enriched in relapsed as well as metastatic tumor specimens. Due to the ubiquity of CIN in cancer cells, it is a potentially way to detect CIN in the cast-off cells from the bile samples for diagnosing and monitoring biliary tract carcinoma patients. BileCAD is a new method to detecting CIN in the DNA sample from patients, including extracting DNA from bile, analyzing DNA by low-coverage whole-genome sequencing, processing the data by bio-information techniques, and finally optimizing the management of biliary tract carcinoma patients.The investigators intended to conduct a prospective study by analyzing bile samples from gallbladder cancers and cholangiocarcinoma patients and control groups that without any tumor in the Bile duct and gallbladder or other organs to compare the specificity and sensitivity of BileCAD test for diagnosing biliary tract carcinoma to other modalities, such as pathological diagnosis. At the same time, the consistency of BileCAD microbial analysis results and clinical microbial culture results was compared, so as to provide more reference for clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* No systemic therapy or biliary tract surgery before the trial.
* Gallstones, bile duct space, obstructive jaundice and other suspected patients with biliary tract carcinoma.
* Male or female patients aged >= 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Age under 18 years.
* Individuals unwilling to sign the consent form or unwilling to provide the medical record.
* Individuals unwilling to participate in this trial.
* Individuals has any active autoimmune disease or history of autoimmune disease.
* Individuals have cardiac clinical symptoms or diseases that are not well controlled.
* Individuals have uncontrolled severe cerebrovascular, pulmonary and other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with biliary tract carcinoma or participants in control group in Taizhou Hospital of Zhejiang Province, Taizhou First People's Hospital, The First Affiliated Hospital of Wenzhou Medical University and Sir Run Run Shaw Hospital from Apr 2023 until the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of bile sample analysis by BileCADanalysis | 12 months
  Number of patients "declared positive" with the BileCAD test among the patients suffered from biliary tract carcinoma.
Specificity of bile sample analysis by BileCADanalysis | 12 months
  Number of patients "declared negative" with the BileCAD test among the patients without cancer.

SECONDARY OUTCOMES:
BileCAD microbial analysis results | 12 months
  Consistency of BileCAD microbial analysis results with clinical microbial culture results
BileCAD analyzed the sensitivity of different types and locations of malignant tumors | 12 months
  The tumors were classified into different types and sites and the sensitivity of BileCAD to different types and sites of malignant tumors was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: fabiao zhang, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University; yunfeng shan, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; ning mu, Principal Investigator — Taizhou First People's Hospital; xiao liang, Principal Investigator — Sir Run Run Shaw Hospital
Locations (4):
- China (4):
  - Sir Run Run Shaw Hospital, School of Medicine，Zhejiang University, Hangzhou, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Richardson TE, Walker JM, Abdullah KG, McBrayer SK, Viapiano MS, Mussa ZM, Tsankova NM, Snuderl M, Hatanpaa KJ. Chromosomal instability in adult-type diffuse gliomas. Acta Neuropathol Commun. 2022 Aug 17;10(1):115. doi: 10.1186/s40478-022-01420-w. PMID 35978439
- [Background] Al-Rawi DH, Bakhoum SF. Chromosomal instability as a source of genomic plasticity. Curr Opin Genet Dev. 2022 Jun;74:101913. doi: 10.1016/j.gde.2022.101913. Epub 2022 May 5. PMID 35526333
- [Background] Bach DH, Zhang W, Sood AK. Chromosomal Instability in Tumor Initiation and Development. Cancer Res. 2019 Aug 15;79(16):3995-4002. doi: 10.1158/0008-5472.CAN-18-3235. Epub 2019 Jul 26. PMID 31350294
- [Background] Liu Y, Yeh MM. Bile duct dysplasia and associated invasive carcinoma: clinicopathological features, diagnosis, and practical challenges. Hum Pathol. 2023 Feb;132:158-168. doi: 10.1016/j.humpath.2022.06.012. Epub 2022 Jun 14. PMID 35714833
- [Background] Onoyama T, Matsumoto K, Koda H, Yamashita T, Kurumi H, Kawata S, Takeda Y, Harada K, Yashima K, Isomoto H. Diagnostic usefulness of KL-6 concentration of bile in biliary tract cancer. Mol Clin Oncol. 2018 Apr;8(4):561-566. doi: 10.3892/mco.2018.1571. Epub 2018 Feb 12. PMID 29541466